CLINICAL TRIAL: NCT01072721
Title: Non Invasive Study of the Hepatic Fibrosis in Paediatrics by the Method of FIBROSCANN.
Brief Title: Non Invasive Study of the Hepatic Fibrosis in Paediatrics by the Method of Study of Pediatric Hepatic Fibrosis
Acronym: PEDISCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P081207; 2009-A00738-49 (Other: AFSSAPS)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cirrhosis; Liver Fibrosis; Portal Hypertension; Cystic Fibrosis; Cholestasis of Parenteral Nutrition
Keywords: Liver; Fibrosis; Elastometry; FIBROSCANN; Children
MeSH Terms: conditions — Fibrosis; Liver Cirrhosis; Hypertension, Portal; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibrosis group (Other): a single arm with the two interventions (elastometry and biopsy)
  Interventions: Other: Elastometry

INTERVENTIONS:
Other: Elastometry — Fibrosis detection with FIBROSCANN

SUMMARY:
Early diagnosis of liver fibrosis is useful for the follow-up and treatment of chronic liver disease. At present, the unique validated method to evaluate the liver fibrosis in children, is the liver biopsy which is an invasive method. If the elastometry method is proved to be a good method to evaluate the fibrosis in children, a numerous liver biopsy could be avoided.

DETAILED DESCRIPTION:
The elastometry method is proved to be efficient for the evaluation of liver fibrosis in adults. But the inter-costal space is too thin in children, and the adult probe could not be used. Recently a special probe adapted to the children have been TECHNICATED. We want to test this specific probe in children. Five French Paediatrics centres will participate to the study. We need 200 children inclusions in 2 years to have a statistically power analysis. Inclusion of each child will be in order to the need of a liver biopsy. Each children included will have an elastometry measure in the same time than the liver biopsy. The fibrosis will be staged by a trained pathologist and scored by METAVIR score witch is the reference. The elastometry measure will be realised by physician with 3 sequential measures in each child. The statistical analysis will be performed by statistician. If elastometry is proved to be an efficient method to evaluate the liver fibrosis in children, a numerous of liver biopsy could be avoided. Because elastometry is a non invasive method it could also be used as follow-up in different categories of children who needs sequential liver biopsy.

ELIGIBILITY:
Inclusion criteria :

* Children age more than 6 months and under 18 years old.
* Children with an hepatic biopsy for any fibrosis hepatitic diseases
* Clinical examination by a physician

Exclusion criteria :

* Children of less than 6 months and more than 18 years old.
* Pregnant women.
* No written informed consent
* No social security

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 264 (Actual)
Dates: Start 2010-01-19 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
To study the diagnosis value of hepatic elasticity measured by FIBROSCANN ® about fibrosis degree in comparison with hepatic biopsy (GOLDSTANDART) in a paediatric hepatic diseases cohort. | until two months

SECONDARY OUTCOMES:
For a better estimation of the fibrosis degree, after measuring the global nature of the liver, by decreasing the sampling bias. | two months
For a best follow-up of the fibrosis to optimize the treatment. | two months

CONTACTS AND LOCATIONS:
Overall Officials: Florence Lacaille, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

REFERENCES:
- [Result] Corpechot C, El Naggar A, Poujol-Robert A, Ziol M, Wendum D, Chazouilleres O, de Ledinghen V, Dhumeaux D, Marcellin P, Beaugrand M, Poupon R. Assessment of biliary fibrosis by transient elastography in patients with PBC and PSC. Hepatology. 2006 May;43(5):1118-24. doi: 10.1002/hep.21151. PMID 16628644
- [Result] Castera L, Vergniol J, Foucher J, Le Bail B, Chanteloup E, Haaser M, Darriet M, Couzigou P, De Ledinghen V. Prospective comparison of transient elastography, Fibrotest, APRI, and liver biopsy for the assessment of fibrosis in chronic hepatitis C. Gastroenterology. 2005 Feb;128(2):343-50. doi: 10.1053/j.gastro.2004.11.018. PMID 15685546
- [Result] Ganne-Carrie N, Ziol M, de Ledinghen V, Douvin C, Marcellin P, Castera L, Dhumeaux D, Trinchet JC, Beaugrand M. Accuracy of liver stiffness measurement for the diagnosis of cirrhosis in patients with chronic liver diseases. Hepatology. 2006 Dec;44(6):1511-7. doi: 10.1002/hep.21420. PMID 17133503
- [Result] de Ledinghen V, Le Bail B, Rebouissoux L, Fournier C, Foucher J, Miette V, Castera L, Sandrin L, Merrouche W, Lavrand F, Lamireau T. Liver stiffness measurement in children using FibroScan: feasibility study and comparison with Fibrotest, aspartate transaminase to platelets ratio index, and liver biopsy. J Pediatr Gastroenterol Nutr. 2007 Oct;45(4):443-50. doi: 10.1097/MPG.0b013e31812e56ff. PMID 18030211